CLINICAL TRIAL: NCT00938431
Title: A Multicenter, Open-Label Study To Investigate The Safety, Tolerability, And Pharmacokinetics Of Lacosamide (LCM) Oral Solution (Syrup) As Adjunctive Therapy In Children With Partial-Onset Seizures
Brief Title: A Multicenter, Open-Label Study To Investigate The Safety And Pharmacokinetics Of Lacosamide In Children With Partial Seizures
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SP0847; 2011-001558-27 (EudraCT Number)
Expanded Access: NCT03559673 (No longer available)
Record Dates: First submitted 2009-07-02; First posted 2009-07-13 (Estimated); Results first posted 2015-12-15 (Estimated); Last update posted 2019-03-19 (Actual); Status verified 2017-07

CONDITIONS: Epilepsy
Keywords: Lacosamide; Vimpat; Children; Epilepsy; Seizures; Anti-epileptic
MeSH Terms: conditions — Epilepsy; Seizures | interventions — Lacosamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Lacosamide - Age 5 - 11 years (Experimental): Cohort 1 (Age 5 - 11 years); up to 8 mg/kg/day
  Interventions: Drug: Lacosamide
- Lacosamide - (Age 12 - 17 years) (Experimental): Cohort 2 (Age 12 - 17 years); 12 mg/kg/day.
  Interventions: Drug: Lacosamide
- Lacosamide (Age 2 - 4 years) (Experimental): Cohort 3 (Age 2 - 4 years); 12 mg/kg/day.
  Interventions: Drug: Lacosamide
- Lacosamide (Age 5 - 11 years) (Experimental): Cohort 4 (Age 5 - 11 years); 12 mg/kg/day.
  Interventions: Drug: Lacosamide
- Lacosamide (Age 1 month - < 2 years) (Experimental): Cohort 5 (Age 1 month to < 2 years); 12 mg/kg/day
  Interventions: Drug: Lacosamide

INTERVENTIONS:
Drug: Lacosamide — Lacosamide oral solution (syrup) 10 mg/mL or 15 mg/mL
  Other Names: Vimpat

SUMMARY:
The purpose of this study was to evaluate the safety and pharmacokinetics of LCM syrup in children ages from 1 month to 17 years with uncontrolled partial seizures when added to 1 to 3 other antiepileptic drugs (AEDs).

DETAILED DESCRIPTION:
Six subjects aged 5-11 (Cohort 1) were initially enrolled at the 8 mg/kg/day dose level. Upon completion of the study for these subjects, pharmacokinetic and safety data were analyzed to determine the target dose for the remaining subjects (either 8, 10 or 12 mg/kg/day). Depending on the selected target dose, four additional age-based cohorts of subjects were to be enrolled. LCM was increased 2 mg/kg/day per week until the target dose or maximum dose able to be tolerated was achieved.

ELIGIBILITY:
Inclusion Criteria:

* Subject is male or female between 1 month and 17 years of age inclusive
* Subject's Body Mass Index (BMI) is within the 5th to 95th percentile for his/her age group
* Subject has a diagnosis of epilepsy with partial-onset seizures
* Subject has been observed to have uncontrolled partial-onset seizures after an adequate course of treatment with at least 2 anti-epileptic drugs (AEDs) (concurrently or sequentially)
* Subject has been observed to have at least 2 countable seizures in the 4-week period prior to Screening
* Subject is on a stable dosage regimen of 1 to 3 AEDs

Exclusion Criteria:

* Subject is currently participating or has participated within the last 2 months in any study of an investigational drug or experimental device
* Subject with seizures that are uncountable due to clustering during the 8-week period prior to study entry
* Subject is on a ketogenic or other specialized diet
* Subject has a history of primary generalized epilepsy
* Subject has a history of status epilepticus within the 6-month period prior to Screening
* Subject is receiving concomitant treatment with felbamate or has received previous felbamate therapy within the last 6 months prior to Screening
* Subject has taken or is currently taking vigabatrin
* Subject is taking monoamine oxidase (MAO) inhibitors or narcotic analgesics
* Subject has a lifetime history of suicide attempt, or has suicidal ideation in the past 6 months

Ages: 1 Month to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 47 (Actual)
Dates: Start 2009-11; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)
Locations (21):
- United States (14):
  - 025, Sacramento, California
  - 002, Washington D.C., District of Columbia
  - 012, Tampa, Florida
  - 019, Wellington, Florida
  - 006, Saint Paul, Minnesota
  - 008, Kansas City, Missouri
  - 015, New Brunswick, New Jersey
  - 005, Durham, North Carolina
  - 001, Philadelphia, Pennsylvania
  - 016, Pittsburgh, Pennsylvania
  - 004, Nashville, Tennessee
  - 026, Austin, Texas
  - 022, Houston, Texas
  - 020, Norfolk, Virginia
- Belgium (3):
  - 201, Brussels
  - 200, Edegem
  - 202, Leuven
- Mexico (4):
  - 101, Culiacán
  - 104, Guadalajara
  - 105, Monterrey
  - 103, San Luis Potosí City

REFERENCES:
- [Result] Winkler J, Schoemaker R, Stockis A. Population Pharmacokinetics of Adjunctive Lacosamide in Pediatric Patients With Epilepsy. J Clin Pharmacol. 2019 Apr;59(4):541-547. doi: 10.1002/jcph.1340. Epub 2018 Nov 14. PMID 30427550
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The SP0847 study began recruitment in October 2009. The study ended in July 2014 with 47 subjects enrolled into the study.
Groups:
- >=1 Month to <4 Years (Safety Set); >=4 Years to <12 Years (Safety Set); >=12 Years to <=17 Years (Safety Set): Subjects were classified as belonging to the age group based on their age at time of enrollment
Period: Overall Study
Arm/Group | >=1 Month to <4 Years (Safety Set) | >=4 Years to <12 Years (Safety Set) | >=12 Years to <=17 Years (Safety Set)
Started | 15 | 23 | 9
Completed | 9 | 14 | 1
Not Completed | 6 | 9 | 8
Not completed — Adverse Event | 5 | 8 | 6
Not completed — Lack of Efficacy | 0 | 1 | 0
Not completed — Did not up titrate to 12 mg kg/day | 1 | 0 | 0
Not completed — Dosing compliance issue | 0 | 0 | 1
Not completed — Reached maximum dose early | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The analysis group for Baseline Characteristics is the Safety Set (SS). The SS is all subjects who signed the informed consent form and took at least 1 dose of Lacosamide (LCM) in SP0847.
Arm/Group | >=1 Month to <4 Years (Safety Set) | >=4 Years to <12 Years (Safety Set) | >=12 Years to <=17 Years (Safety Set) | Total Title
Number analyzed (Participants) | 15 | 23 | 9 | 47
Age, Continuous [Mean (Standard Deviation); unit: years]
  Age (years) | 1.58 (1.02) | 7.41 (2.44) | 15.15 (1.50) | 7.03 (5.12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 9 | 5 | 24
  Male | 5 | 14 | 4 | 23
Weight [Mean (Standard Deviation); unit: kilograms] | 9.90 (3.31) | 26.73 (10.20) | 54.10 (10.49) | 26.60 (17.64)
Height [Mean (Standard Deviation); unit: centimeters] | 79.64 (11.22) | 121.81 (14.86) | 158.93 (11.43) | 115.46 (31.23)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 15.27 (2.33) | 17.39 (2.68) | 21.38 (3.12) | 17.48 (3.37)
Racial Group [Number; unit: participants]
  Asian | 1 | 1 | 0 | 2
  Black | 0 | 4 | 3 | 7
  White | 7 | 18 | 5 | 30
  Other/ Mixed | 7 | 0 | 1 | 8
Ethnicity [Number; unit: participants]
  Hispanic or Latino | 11 | 7 | 3 | 21
  Not Hispanic or Latino | 4 | 16 | 6 | 26

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects That Report at Least One Treatment-emergent Adverse Event During the Study (Approximately 13 Weeks)
Time Frame: 13 weeks
Population: The analysis consists of the Safety Set (SS), which is all subjects who signed the informed consent form and took at least 1 dose of Lacosamide (LCM) in SP0847.
Measure: Number; unit: participants
Arm/Group | >=1 Month to <4 Years (Safety Set) | >=4 Years to <12 Years (Safety Set) | >=12 Years to <=17 Years (Safety Set)
Number analyzed (Participants) | 15 | 23 | 9
participants | 14 | 19 | 9

2. Secondary Outcome: Change in Seizure Frequency From Baseline to End of Treatment
Time Frame: From Baseline to End of Treatment (approximately 13 weeks)
Population: This analysis consists of the Full Analysis Set, which is all subjects from the Safety Set who have at least 1 post-Baseline seizure diary day with available data during the SP0847 study.
Measure: Mean (Standard Deviation); unit: percentage change
Groups:
- >=1 Month to <4 Years (Full Analysis Set); >=4 Years to <12 Years (Full Analysis Set); >=12 Years to <=17 Years (Full Analysis Set): Subjects were classified as belonging to the age group based on their age at time of enrollment
Arm/Group | >=1 Month to <4 Years (Full Analysis Set) | >=4 Years to <12 Years (Full Analysis Set) | >=12 Years to <=17 Years (Full Analysis Set)
Number analyzed (Participants) | 14 | 23 | 9
percentage change | 18.94 (111.44) | 18.38 (88.16) | 34.59 (92.45)

3. Secondary Outcome: Caregiver Global Impression of Change Score at Visit 5 (Day 27/28) or Early Termination
Description: For the assessment of the Caregiver Global Impression of Change, the caregiver (including parent/legal guardian) provided his/her assessment of the subject's clinical status, compared to Baseline (Visit 1), including an evaluation of seizure frequency and intensity, the occurrence of Adverse Events (AEs), and subject's functional status.
  The caregiver will be asked to check the number that best describes the subject's condition over the past 4 weeks compared to Baseline:
  1. Very much improved
  2. Much improved
  3. Minimally improved
  4. No change
  5. Minimally worse
  6. Much worse
  7. Very much worse
Time Frame: Visit 5 (Day 27/28) or Early Termination
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | >=1 Month to <4 Years (Full Analysis Set) | >=4 Years to <12 Years (Full Analysis Set) | >=12 Years to <=17 Years (Full Analysis Set)
Number analyzed (Participants) | 14 | 23 | 9
Participants
  Very Much Improved | 3 | 2 | 0
  Much Improved | 7 | 8 | 4
  Minimally Improved | 3 | 8 | 3
  No Change | 0 | 2 | 1
  Miniamally Worse | 0 | 1 | 0
  Much Worse | 0 | 2 | 0
  No data available | 1 | 0 | 1

4. Secondary Outcome: Clinical Global Impression of Change Score at Visit 5 (Day 27/28) or Early Termination
Description: For assessment of the Clinical Global Impression of Change, the investigator provided his/her assessment of the subject's clinical status, compared to Baseline (Visit 1), including an evaluation of seizure frequency and intensity, the occurrence of AEs, and subject's functional status.
  The investigator will be asked to check the number that best describes the subject's condition over the past 4 weeks compared to Baseline:
  1. Very much improved
  2. Much improved
  3. Minimally improved
  4. No Change
  5. Minimally worse
  6. Much worse
  7. Very much worse
Time Frame: Visit 5 (Day 27/28) or Early Termination
Population: This analysis consists of the Full Analysis Set, which is all subjects from the Safety Set who have at least 1 post-Baseline seizure diary day with available data during the SP0847 study.
  For one subject in the age group >=12 years to <=17 years no data is available.
Measure: Number; unit: Participants
Arm/Group | >=1 Month to <4 Years (Full Analysis Set) | >=4 Years to <12 Years (Full Analysis Set) | >=12 Years to <=17 Years (Full Analysis Set)
Number analyzed (Participants) | 14 | 23 | 9
Participants
  Very Much Improved | 2 | 2 | 0
  Much Improved | 6 | 7 | 7
  Minimally Improved | 4 | 9 | 1
  No Change | 1 | 2 | 0
  Minimally Worse | 0 | 3 | 0
  Much Worse | 1 | 0 | 0
  No data available | 0 | 0 | 1

5. Secondary Outcome: Plasma Ctrough Values for Lacosamide at Day 7
Description: During SP0847, the time points for collection of blood samples for plasma concentration analysis varied per enrollment cohort. To provide a standard summary of this information, we present the mean plasma trough concentrations (Ctrough). Ctrough levels represent the lowest level of LCM that was present in the subject with measurement taken pre-dose before the next scheduled dose of LCM.
  The blood sample for plasma concentration schedule varied per enrollment cohort and with protocol amendments. A PK sample was not required for a subject to be in the included in the SS although all subjects did have at least one PK sample taken during SP0847. Therefore the number of subjects presented for the PK assessments is based on the subjects in the SS who attended the respective visits and had PK concentration data at the respective time point.
Time Frame: Day 7
Population: The analysis consists of the Safety Set, which is all subjects who signed the informed consent form and took at least 1 dose of LCM in SP0847.
  The number of subjects presented for the PK assessments is based on the subjects in the SS who attended the respective visits and had PK concentration data at the respective time point.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Groups:
- All Subjects (Safety Set): All subjects from >=1 month to <=17 years
Arm/Group | All Subjects (Safety Set)
Number analyzed (Participants) | 45
μg/mL | 839.9 (64.1)

6. Secondary Outcome: Plasma Ctrough Values for Lacosamide at Day 28
Description: as for outcome 5
Time Frame: Day 28
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | All Subjects (Safety Set)
Number analyzed (Participants) | 6
μg/mL | 3886.0 (70.2)

7. Secondary Outcome: Plasma Ctrough Values for Lacosamide at Day 35
Description: as for outcome 5
Time Frame: Day 35
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | All Subjects (Safety Set)
Number analyzed (Participants) | 5
μg/mL | 4033.8 (52.5)

8. Secondary Outcome: Plasma Ctrough Values for Lacosamide at Day 42
Description: as for outcome 5
Time Frame: Day 42
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | All Subjects (Safety Set)
Number analyzed (Participants) | 14
μg/mL | 4169.5 (73.3)

9. Secondary Outcome: Plasma Ctrough Values for SPM 12809 at Day 7
Description: SPM 12809 is major metabolite of LCM and is known as O-desmethyl-lacosamide. During SP0847, the time points for collection of blood samples for plasma concentration analysis varied per enrollment cohort. To provide a standard summary of this information, we present the mean plasma trough concentrations (Ctrough). Ctrough levels represent the lowest level of LCM that was present in the subject with measurement taken pre-dose before the next scheduled dose of LCM.
  The blood sample for plasma concentration schedule varied per enrollment cohort and with protocol amendments. A PK sample was not required for a subject to be in the included in the SS although all subjects did have at least one PK sample taken during SP0847. Therefore the number of subjects presented for the PK assessments is based on the subjects in the SS who attended the respective visits and had PK concentration data at the respective time point.
Time Frame: Day 7
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | All Subjects (Safety Set)
Number analyzed (Participants) | 45
μg/mL | 258.4 (44.6)

10. Secondary Outcome: Plasma Ctrough Values for SPM 12809 at Day 28
Description: as for outcome 9
Time Frame: Day 28
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | All Subjects (Safety Set)
Number analyzed (Participants) | 6
μg/mL | 754.9 (21.1)

11. Secondary Outcome: Plasma Ctrough Values for SPM 12809 at Day 35
Description: as for outcome 9
Time Frame: Day 35
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | All Subjects (Safety Set)
Number analyzed (Participants) | 5
μg/mL | 955.1 (24.7)

12. Secondary Outcome: Plasma Ctrough Values for SPM 12809 at Day 42
Description: as for outcome 9
Time Frame: Day 42
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | All Subjects (Safety Set)
Number analyzed (Participants) | 14
μg/mL | 1725.8 (39.4)

ADVERSE EVENTS:
Time Frame: Adverse Events (AE) and Serious Adverse Events (SAE) were recorded for the duration of the study (November 2009 - July 2014). The analysis group for AEs and SAEs was the Safety Set.
Description: The Safety Set comprised of all subjects who signed the informed consent form and took at least 1 dose of Lacosamide in SP0847.
Arm/Group | >=1 Month to <4 Years (Safety Set) | >=4 Years to <12 Years (Safety Set) | >=12 Years to <=17 Years (Safety Set)
Serious Adverse Events (participants affected / at risk) | 3/15 | 3/23 | 0/9
Other Adverse Events (participants affected / at risk) | 11/15 | 16/23 | 7/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | >=1 Month to <4 Years (Safety Set) (N=15) | >=4 Years to <12 Years (Safety Set) (N=23) | >=12 Years to <=17 Years (Safety Set) (N=9)
Gastrointestinal inflammation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pneumonia viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Status epilepticus (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | >=1 Month to <4 Years (Safety Set) (N=15) | >=4 Years to <12 Years (Safety Set) (N=23) | >=12 Years to <=17 Years (Safety Set) (N=9)
Vomiting (Gastrointestinal disorders) | 1 (3) | 7 (7) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 4 (7) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
Irritability (General disorders) | 3 (3) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 2 (2) | 3 (4) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 2 (2) | 1 (1)
Otitis media (Infections and infestations) | 0 (0) | 3 (3) | 0 (0)
Pharyngotonsillitis (Infections and infestations) | 3 (3) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 2 (2) | 3 (3) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 3 (4) | 2 (2)
Balance disorder (Nervous system disorders) | 0 (0) | 1 (2) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
UCB has > 60 but <= 180 days to review results communications prior to public release and may delete information that is confidential and compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that the results shall be published regardless of outcome.